CLINICAL TRIAL: NCT02464072
Title: Randomized Clinical Trial of Subtotal Parathyroidectomy or Total Parathyroidectomy With Immediate Heterotopic Autograft in Chronic Renal Disease Patients Stage V Under Dialysis
Brief Title: Subtotal Parathyroidectomy or Total Parathyroidectomy With Autograft in Chronic Kidney Disease Patients Under Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Sergio Arap, Attending Physcian, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 00828412.8.0000.0068
Record Dates: First submitted 2015-05-18; First posted 2015-06-08 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Hyperparathyroidism, Secondary
Keywords: Parathyroidectomy; Renal Insufficiency, Chronic
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subtotal Parathyroidectomy (Experimental): Patients will be submitted to subtotal parathyroidectomy. The intention is to leave a parathyroid remanent equivalent to two normal parathyroid glands in situ. The type of the operation is the intervention. No drugs or devices are tested.
  Interventions: Procedure: Subtotal Parathyroidectomy
- Total Parathyroidectomy + 45 autografts (Active Comparator): Patients will be submitted to a total parathyroidectomy and 45 fragments of parathyroid tissue are grafted in the forearm. This is the current standard treatment at the institution for severe secondary hyperparathyroidism.The type of operation is the intervention itself. No new device or drug is involved.
  Interventions: Procedure: Total Parathyroidectomy + 45 autografts
- Total Parathyroidectomy + 90 autografts (Experimental): Patients will be submitted to a total parathyroidectomy and 90 fragments of parathyroid tissue are grafted in the forearm. The type of operation is the intervention. No new device or drug is involved. .
  Interventions: Procedure: Total Parathyroidectomy + 90 autografts

INTERVENTIONS:
Procedure: Subtotal Parathyroidectomy — Subtotal parathyroid resection leaving the estimated mass of two normal parathyroid glands in situ. The type of operation is the intervention. No new device or drug is involved.
  Arms: Subtotal Parathyroidectomy
Procedure: Total Parathyroidectomy + 45 autografts — Immediate autograft of 45 fragments of parathyroid tissue, after a total parathyroidectomy.This type of operation is the standard intervention at the institution at the moment. No new device or drug is involved.
  Arms: Total Parathyroidectomy + 45 autografts
Procedure: Total Parathyroidectomy + 90 autografts — Immediate autograft of 90 fragments of parathyroid tissue, after a total parathyroidectomy.The type of operation is the intervention. No new device or drug is involved.
  Arms: Total Parathyroidectomy + 90 autografts

SUMMARY:
This study evaluates the metabolic and clinical results of two well recognized and accepted surgical techniques in the management of severe hyperparathyroidism in patients under regular dialysis treatment.

DETAILED DESCRIPTION:
Prospective randomized trial in the surgical management of severe hyperparathyroidism of chronic kidney disease stage V under dialysis. Patients will be randomized and they will be submitted to subtotal parathyroidectomy or total parathyroidectomy with immediate heterotopic autograft of 45 or 90 fragments of parathyroid tissue.

ELIGIBILITY:
Inclusion Criteria:

* Stage V Chronic Kidney Disease patients under regular dialysis treatment with severe hyperparathyroidism requiring parathyroidectomy

Exclusion Criteria:

* patients refusing to participate in the study (they will receive standard surgery),
* patients unable to attend regular follow up consultations,
* patients with a successful kidney transplant at the moment of parathyroidectomy,
* patients submitted to any previous surgery of the thyroid or parathyroid,
* patients with chronic kidney disease but not under dialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Survival | From the time of the operation until 5 years after intervention or death if it occurs before 5 years of follow up
  Five years survival after parathyroidectomy in an intention to treat analysis

SECONDARY OUTCOMES:
Metabolic Outcome 1: Serum Calcium (mg/dL) | 1 to 60 months after intervention, Samples are taken according to regular follow up
  postoperative calcium levels. Below, Above or in the normal range for the method. Analysis will include samples taken close to 1, 3, 6, 12, 24, 36, 48 and 60 months after the operation.
Metabolic Outcome 2 : Serum Phosphorus (mg/dL) | 1 to 60 months after intervention, Samples are taken according to regular follow up
  postoperative phosphorus levels. Below, above or the normal range for the method employed. Analysis will include samples taken close to 1, 3, 6, 12, 24, 36, 48 and 60 months after the operation.
Metabolic Outcome 3: Serum Alkaline Phosphatase (IU) | 1 to 60 months after intervention, Samples are taken according to regular follow up
  postoperative alkaline phosphatase levels. Above or in the normal range, according to the method in use. Analysis will include samples taken close to 1, 3, 6, 12, 24, 36, 48 and 60 months after the operation.
Metabolic Outcome 4: Serum Parathormone (pg/mL) | 1 to 60 months after intervention, Samples are taken according to regular follow up
  postoperative parathormone levels. Below, Above or in the target levels proposed by the National Kidney Foundation, and by the Kidney Disease Improving Global Outcomes (KDIGO). Analysis will include samples taken close to 1, 3, 6, 12, 24, 36, 48 and 60 months after the operation.
Drug Requirement 1: Elemental Calcium Intake (g/day) | 1 to 60 months after intervention, according to the dose prescibed in different periods.
  The calcium supplement intake (in grams of elemental calcium per day) of the patients after the intervention. Analysis will include first week, then 1, 3, 6, 12, 24,36, 48, 60 months after the intervention.
Drug Requirement 2 Calcitriol intake (micrograms/day) | 1 to 60 months after intervention, according to the dose prescibed in different periods
  calcitriol or other vitamin D analogue intake (in micrograms per day) after the intervention. Analysis will include first week, then 1, 3, 6, 12, 24,36, 48, 60 months after the intervention.
Drug Requirement 3: Sevelamer (mg/day) | 1 to 60 months after intervention, according to the dose prescibed in different periods
  The quantity of phosphorus binding drugs, in special Sevelamer prescribed in milligrams after the intervention. Analysis will include 1, 3, 6, 12, 24,36, 48, 60 months after the operation.
Drug Requirement 4: Calcimimetics (mg/day) | 1 to 60 months after intervention, according to the dose prescibed in different periods
  The amount of Calcimimetics, in special Cinacalcet im milligrams per day prescribed after the intervention. Analysis will include 1, 3, 6, 12, 24,36, 48, 60 months after the intervention.
Clinical Outcome 1: Bone Pain in the VAS | Pre-operative (up to one week before the procedure) until 60 months after intervention
  Bone pain measured by the Visual Analogic Pain Scale up to one week before the intervention and up to one week after the procedure, and then at regular follow up. Analysis will concentrate on preoperative (up to one week before), postoperative up to one week, 6,12, 24, 36, 48 and 60 months after the intervention.
Clinical Outcome 2: Postoperative Skeletal Disease (Fractures/Brown tumor) | 1 to 60 months after intervention
  skeletal disease is defined as the occurrence of a fracture or the developement brown tumor (osteoclastomas) after the intervention, detected clinically or by any clinically oriented radiography ordered by the attending physician in routine follow up or in any emergency setting.
Clinical Outcome 3: Quality of Life in the SF-36 Questionnaire | Preoperative (up to three days before the intervention) and until 60 months after intervention
  quality of life up to one week before the intervention and after the operation at one week, 6 , 12, 24, 36, 48 and 60 months, measured by the Short form 36 questionnaire (SF-36) validated to the cultural and language of the country.
Clinical Outcome 4: Additional Operation (Reoperation in Recurrent/Persistent Disease) | 1 to 60 months after intervention
  the necessity of reoperative procedures due to recurrence or persistence of severe hyperparathyroidism, as defined by the attending physician during regular follow up
Morbidity of the surgical procedures | intra-operative to 60 months
  After any interventions (initial operation or reoperative interventions necessary in the follow up), it will be actively searched for the occurrence of dysphonia (and its cause according to laryngoscopy), wound infection (clinical signs as red skin, pain, secretion, fever and laboratory evidence), and neck haematoma (large neck blood clots requiring operation)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio S Arap, M.D., Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filho WA, van der Plas WY, Brescia MDG, Nascimento CP Jr, Goldenstein PT, Neto LMM, Arap SS, Custodio MR, Bueno RO, Moyses RMA, Jorgetti V, Kruijf S, Montenegro FLM. Quality of life after surgery in secondary hyperparathyroidism, comparing subtotal parathyroidectomy with total parathyroidectomy with immediate parathyroid autograft: Prospective randomized trial. Surgery. 2018 Nov;164(5):978-985. doi: 10.1016/j.surg.2018.06.032. Epub 2018 Aug 3. PMID 30082137
- [Background] Albuquerque RFC, Carbonara CEM, Martin RCT, Dos Reis LM, do Nascimento CP Junior, Arap SS, Moyses RMA, Jorgetti V, Montenegro FLM, de Oliveira RB. Parathyroidectomy in patients with chronic kidney disease: Impacts of different techniques on the biochemical and clinical evolution of secondary hyperparathyroidism. Surgery. 2018 Feb;163(2):381-387. doi: 10.1016/j.surg.2017.09.005. Epub 2017 Nov 13. PMID 29146232
- [Background] Silveira AA, Brescia MDG, do Nascimento CP Jr, Arap SS, Montenegro FLM. Critical analysis of the intraoperative parathyroid hormone decrease during parathyroidectomy for secondary and tertiary hyperparathyroidism. Surgery. 2020 Dec;168(6):1079-1085. doi: 10.1016/j.surg.2020.06.043. Epub 2020 Aug 15. PMID 32811697
- [Derived] Pereira GMD, Liao M, Arap SS, Magnabosco FF, Brescia MDG, Moyses RMA, Custodio MR, Jorgetti V, Kowalski LP, Montenegro FLM. Parathyroidectomy reduces the costs of medication in patients with secondary hyperparathyroidism. Clinics (Sao Paulo). 2024 Sep 15;79:100484. doi: 10.1016/j.clinsp.2024.100484. eCollection 2024. PMID 39284277
- [Derived] Silveira AA, Brescia MDG, Nascimento CPD Jr, Arap SS, Montenegro FLM. Delayed sampling of intraoperative parathormone may be unnecessary during parathyroidectomy in kidney-transplanted and dialysis patients. J Bras Nefrol. 2021 Apr-Jun;43(2):228-235. doi: 10.1590/2175-8239-JBN-2020-0108. PMID 33475675